CLINICAL TRIAL: NCT07389369
Title: Comparison of International Physical Activity Questionnaire Levels and Smartwatch-Measured Physical Activity Levels in University Students
Brief Title: Comparison of a Subjective Questionnare With Daily Step Count
Status: Completed | Type: Observational
Sponsor: Istanbul Aydın University (Other)
Responsible Party: Principal Investigator, İoakim İpseftel, Assistant Professor at Health Sciences Faculty Physiotherapy and Rehabilitation Department, Istanbul Aydın University
Other Study IDs: İAU-SBF-FTR-İİ-01
Record Dates: First submitted 2026-01-16; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Physical Activities; Daily Activities
Keywords: Physical Activity; Daily Step Counts; Accelerometry; Questionnaire; Sleep Quality
MeSH Terms: conditions — Motor Activity; Sleep Initiation and Maintenance Disorders | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- university students: The university students who are actively attending classes.
  Interventions: Device: Daily step counting with a smartwatch; Other: Questionnaire

INTERVENTIONS:
Device: Daily step counting with a smartwatch — daily step count measurement with a smartwatch
Other: Questionnaire — This questionnaire provides a description of the weekly level of activities.

SUMMARY:
The aim of this study is to explore the correlation between the physical activity levels of university students, as measured by the International Physical Activity Questionnaire-Short Form (IPAQ-SF)(SUBJECTİVE DATA) and their daily step count recorded by Apple smartwatches (OBJECTİVE DATA).

DETAILED DESCRIPTION:
Healthy individuals can monitor their physical activity, sleep quality, and vital signs through smartwatches and mobile applications. Tracking daily step counts via smartwatches helps individuals observe their physical activity levels and boost their motivation. This study aims to explore the correlation between the physical activity levels of university students, as measured by the International Physical Activity Questionnaire-Short Form (IPAQ-SF), and their daily step count recorded by Apple smartwatches. Moreover, this investigation examined the feasibility of employing daily step count -a more objective measure-instead of the categorical data generally utilized in evaluating IPAQ scores in existing literature. It is suggested that this methodology may mitigate subjectivity and advance future research efforts. Additionally, the relationship between the students' physical activity levels and sleep quality was evaluated. The research involved 102 volunteer students from Istanbul Aydın University. Participants' average daily step counts were documented from their smartwatches over a week, followed by the completion of IPAQ-SF and the Pittsburgh Sleep Quality Index (PSQI).

ELIGIBILITY:
Inclusion criteria:

* being a student at Istanbul Aydın University,
* age between 18 and 28 years,
* regular use of an Apple Watch,
* voluntary participation.

Exclusion criteria:

* presence of chronic diseases,
* physical or mental disabilities that could potentially affect physical activity levels,
* being a professional athlete.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 120 university students who take classes
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Correlation of IPAQ and daily step counts of university students | one week for each participant
  This study aims to explore the correlation between the physical activity levels of university students, as measured by the International Physical Activity Questionnaire-Short Form (IPAQ-SF)(SUBJECTİVE DATA) and their daily step count recorded by Apple smartwatches (OBJECTİVE DATA).

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul Aydin University, Istanbul, Bakırköy, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No